CLINICAL TRIAL: NCT05262816
Title: Urodynamic Analysis of the Effect of Electroacupuncture at Different Acupoints on Bladder Function After Spinal Cord Injury
Brief Title: Effect of Electroacupuncture at Different Acupoints on Bladder Function After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2021-15-103
Record Dates: First submitted 2021-09-07; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Neurogenic Bladder
Keywords: Electroacupuncture; Neurogenic Bladder; Spinal Cord Injury
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sanyinjiao group (Experimental): Perpendicular insertion about 0.8-1.2cun at bilateral sanyinjiao(SP6) acupoint.Then,bilateral SP6 were connected with Electronic Acupuncture Treatment Instrument (KWD-808-I,Yingdi, China). The frequency of the pulse was 20 Hz with a pulse duration of 200 us.Intensity of stimulus was depending on patient's tolerance.
  Interventions: Other: electroacupuncture
- guanyuan group (Active Comparator): Perpendicular insertion about 0.8-1.2cun at bilateral Guanyuan(CV4), Zhongji (CV3) acupoints.Then,the two acupoints were connected with Electronic Acupuncture Treatment Instrument (KWD-808-I,Yingdi, China). The frequency of the pulse was 20 Hz with a pulse duration of 200 us.Intensity of stimulus was depending on patient's tolerance.
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — electroacupuncture at Sanyinjiao (SP6)

SUMMARY:
Neurogenic bladder after spinal cord injury can be divided into detrusor hyperreflexia and detrusor non reflexia. Acupuncture is recognized as a safe and effective treatment. The most commonly used acupoints are Guanyuan, Zhongji and Sanyinjiao. The purpose of this study is to clarify the therapeutic effects of different acupoints on different types of bladder. Main process: routine urodynamic examination was performed first, and then electroacupuncture was given to Guanyuan, Zhongji and Sanyinjiao points respectively, and urodynamic examination was performed again to observe the effect of Electroacupuncture on urodynamic parameters in real time.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with traumatic suprasacral SCI.
* the period of the spinal shock has passed.
* patients with voiding dysfunction after SCI.
* patients had stable condition, and suitable for treatment.
* agreed to engage in our study and sign the informed consent.

Exclusion Criteria:

* Patients with severe primary diseases such as heart, liver, kidney, hematopoietic system, endocrine system and psychosis.
* dysuria caused by non spinal cord injury, such as prostatic hypertrophy, urethral obstruction, operation.
* Patients who have already taken cystostomy and sacral electrode implantation.
* Patients with urinary tract infection.
* Autonomic hyperreflexes were obvious.
* Unable to cooperate with the healer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Perianal surface electromyography | Procedure (While doing acupuncture )
  Perianal surface electromyography
detrusor overactivity (DO) | Procedure (While doing acupuncture )
  detrusor overactivity in milliliter,one of the urodynamic parameters
bladder compliance (BC) | Procedure (While doing acupuncture )
  bladder compliance in ml/cmH2O,one of the urodynamic parameters
maximum cystometric capacity (MCC) | Procedure (While doing acupuncture )
  maximum cystometric capacity in milliliter,one of the urodynamic parameters
maximum urinary flow rate (Qmax) | Procedure (While doing acupuncture )
  maximum urinary flow rate in milliliter/second,one of the urodynamic parameters
maximum detrusor pressure | Procedure (While doing acupuncture )
  maximum detrusor pressure at filling stage and voiding stage

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China